CLINICAL TRIAL: NCT05672784
Title: Genicular Nerve Block Versus Its Combination With Infiltration Between Popliteal Artery and Capsule of Posterior Knee for Enhanced Recovery After Total Knee Arthroplasty
Brief Title: Genicular Nerve Block Versus Its Combination With Infiltration Between Popliteal Artery and Capsule of Posterior Knee
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba M Fathi, Dr. Heba M Fathi, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9577/19-9-2022
Record Dates: First submitted 2022-11-05; First posted 2023-01-05 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain
Keywords: genicular ,IPACK, total knee
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Meloxicam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- C group (Active Comparator): the patients will take standard analgesia ( meloxicam (15 mg) once a day + paracetamol 1gm /3 times a day). ,with no nerve block
  Interventions: Drug: standard analgesia (paracetamol and meloxicam)
- G group (Active Comparator): the patients will take standard analgesia plus GNB
  Interventions: Procedure: GNB plus standard analgesia; Drug: standard analgesia (paracetamol and meloxicam)
- GI group (Active Comparator): the patients will take standard analgesia plus GNB plus IPACK
  Interventions: Procedure: GNB plus IPACK block plus standard analgesia; Drug: standard analgesia (paracetamol and meloxicam)

INTERVENTIONS:
Procedure: GNB plus standard analgesia — When patients are in supine position with a pillow under the popliteal fossa, we will target points next to superior medial, superior lateral, and inferior medial genicular arteries to block the superior medial, superior lateral, and inferior medial branches of genicular nerve. For identification, we will use color Doppler near the periosteal areas (the junctions of the epicondyle with the shafts of the femur and tibia, accordingly). using a 12 MHz linear transducer (XarioTM SSA-660A, Toshiba Medical Systems Corporation, Otawara, Japan) positioned parallel to the shaft of the long bones in the legs, the needle will be inserted ( in plane technique in the long-axis view) and a 2.5 mL of bupivacaine (5%) will be injected at each target points.standard analgesia will be given post-operativelly (paracetamol 1 gm/ three times a daily and meloxicam (15 mg)once a day)
  Other Names: genicular block and standard analgesia
  Arms: G group
Procedure: GNB plus IPACK block plus standard analgesia — IPACK block will be done when the patients in supine position with the knee flexed in 45 degree. using a low frequency transducer at a depth of 3.5-4 cm positioned transversely, 2-3 cm above the patella and over the medial aspect of the knee, we will identify the distal part of the shaft of the femur and the popliteal artery with sliding the transducer proximally and distally (If the two femoral condyles appear first, proximal sliding of the probe, so the humps of the femoral condyles will disappeared and the flat metaphysis will appeared). With advancement of the needle in plane toward the space between the popliteal artery and the femur, 15 ml of bupivacaine 0.5% will be injected. The genicular nerve block will be done as in group G and standard analgesia will be given post-operative as in group G
  Other Names: genicular bock and IPACK block and standard analgesia
  Arms: GI group
Drug: standard analgesia (paracetamol and meloxicam) — (paracetamol 1 gm 3 times a daily and meloxicam (15 mg) once aday.
  Other Names: standard analgesia with no nerve block

SUMMARY:
Comparison of the analgesic and physical recovery effect of genicular nerve block (GNB) alone and (GNB + infiltration between popliteal artery and posterior capsule of the knee (IPACK) in patients undergoing total knee replacement

DETAILED DESCRIPTION:
Comparison of preemptive analgesia of (GNB) with (GNB+ IPACK) on postoperative pain control and recovery of knee physical activity in patient undergoing total knee replacement.

ELIGIBILITY:
Inclusion criteria:

* Adult patients aged between 21 to 60 years
* undergoing primary unilateral elective total knee arthroplasty under spinal anesthesia
* Having informed consents
* patients with physical status ASA I & II
* both genders
* body mass index less than 40 kg/m2.

Exclusion criteria

* patients with Peripheral vascular disease
* patients with history of allergy to local anesthesia or opioid analgesia,
* those on anti-platelet, anticoagulant or B blocker drugs
* Patients with acute decompensated heart failure
* Patients with hypertension
* Patients with heart block
* Patients with coronary disease
* Patients with bronchial asthma
* Patients with bleeding disorders
* Patients with compromised renal or hepatic function
* pregnant female.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-11-05 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
2 hours visual analogue scale | at 2 hour postoperative.
  pain intensity at rest and with motion using visual analogue scale from " horizontal line of 10-cm long with two ends, one end indicate no pain 0 and the other end indicate worst pain 10".
4 hours visual analogue score | at 4 hours postoperative
  pain intensity at rest and with motion using visual analogue scale from " horizontal line of 10-cm long with two ends, one end indicate no pain 0 and the other end indicate worst pain 10".
6 hours visual analogue score | at 6 hours postoperative
  pain intensity at rest and with motion using visual analogue scale from " horizontal line of 10-cm long with two ends, one end indicate no pain 0 and the other end indicate worst pain 10".
8 hours visual analogue score | at 8 hours postopertaive
  pain intensity at rest and with motion using visual analogue scale from " horizontal line of 10-cm long with two ends, one end indicate no pain 0 and the other end indicate worst pain 10".
12 hours visual analogue score | at 12 hours postoperative
  pain intensity at rest and with motion using visual analogue scale from " horizontal line of 10-cm long with two ends, one end indicate no pain 0 and the other end indicate worst pain 10".
18 hours visual analogue score | at 18 hours postoperative
  pain intensity at rest and with motion using visual analogue scale from " horizontal line of 10-cm long with two ends, one end indicate no pain 0 and the other end indicate worst pain 10".
24 hours visual analogue score | at 24 hours postoperative
  pain intensity at rest and with motion using visual analogue scale from " horizontal line of 10-cm long with two ends, one end indicate no pain 0 and the other end indicate worst pain 10".

SECONDARY OUTCOMES:
• Time of performance of block | from putting of U.S probe till the end of block procedure
  defined as time from putting of U.S probe till the end of block procedure.
• Total morphine consumption | at 24 hours post-operatively
  Total morphine consumption
•incidence of Anticipated side effect | at 24,48 hours postoperative
  nausea, vomiting, itching, hemorrhage, bradycardia and hypotension.
degree of maximum active flexion and extension of the knee | at 24 hours post operative
  the angle of maximum active flexion and extension of the knee
walk test | at 24 hours post operative
  walking distance in meters that patients can wake during 2 min
holding quadriceps muscle | at 24 hours post operative
  number of patients capable to hold quadriceps muscle more than 5 seconds.
time up and go (TUG) | at 24 hours post operative
  the time required for the patient to stand up from a standard-height armchair, walk 3 meters, turn, walk back to the chair, and sit down

CONTACTS AND LOCATIONS:
Locations (1):
- Heba M Fathi, Zagazig, Egypt

REFERENCES:
- [Derived] Fathi HM, Fahmy AM, Shaker MA, Kamel AAF. Comparison of genicular nerve block and its combination with IPACK block for analgesia and recovery after total knee arthroplasty: a randomized trial. BMC Anesthesiol. 2025 Nov 29;25(1):601. doi: 10.1186/s12871-025-03408-0. PMID 41318369